CLINICAL TRIAL: NCT05671198
Title: Ultrasound of the Diaphragm As Physiological Biomarker in Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Sonographic Diaphragm Function in AECOPD
Acronym: UNDATED
Status: Recruiting | Type: Observational
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Wytze de Boer, Coördinating Investigator, Isala
Other Study IDs: Diaphragm 002
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Copd
Keywords: diaphragm; COPD; thoracic ultrasound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Ultrasound of the diaphragm — Sonographic parameters of the diaphragm:
  * Thickening Fraction (TF); (Diaphragm thickness end-inspiration- Diaphragm thickness end-expiration) / Diaphragm thickness end-expiration. (continuous variable).
  * Diaphragm end-expiratory thickness: Diaphragm thickness at end-expiration (continuous variable)
  * Diaphragm excursion (DE): diaphragm inspiratory amplitude during deep breathing (continuous variable).

SUMMARY:
The study will be conducted as a single-center, prospective cohort study. The primary objective of this study is to investigate the responsiveness of sonographic parameters of diaphragm to detect change in Borg score for dyspnea during hospitalisation for AECOPD without respiratory acidosis.

DETAILED DESCRIPTION:
To investigate the responsiveness of sonographic parameters to detect change in Borg score for dyspnea during hospitalisation for AECOPD without respiratory acidosis, we propose a prospective cohort design.

After inclusion, participants will have assessment of diaphragm function (excursion, thickness, thickening fraction) using ultrasound within 48 hours of admission to the emergency ward, striving to assessment within 24 hours of admission. Additionally, dyspnea grade will be assessed using validated questionnaires.

Further diagnostic work-up and treatment for AECOPD is performed at the discretion of the treating physician.

Both ultrasound measurements and dyspnea grade questionnaires will be repeated when the participant is reported suitable for hospital discharge by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation primarily because of severe acute exacerbation of COPD
* COPD, according to GOLD 2018 definition
* Post-bronchodilator FEV1/FVC < 0,70 and FEV1% < 80%pred. within last 5 years

Exclusion Criteria:

* Respiratory acidosis (pH < 7.35 ánd PaCO2 > 6 kPA)
* Need for (non-)invasive ventilation based on other criteria (e.g. severe hypoxia) upon presentation.
* Established diagnosis of diaphragm diaphragm paralysis.
* Inability for diaphragm imaging (e.g. mechanical ventilation, or unable to follow vocal instructions).
* Those not able or unwilling to give written informed consent.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our population consists of 18-years or older patients who are hospitalised primarily due to AECOPD without respiratory acidosis.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
- To investigate the responsiveness of sonographic parameters to detect change in Borg score for dyspnea during hospitalisation for AECOPD without respiratory acidosis. | from admission till hospital discharge (expected median of 5 days based on experience)
  Correlation between:
  * Change in Borg score for dyspnea; defined as score at discharge minus score at admission
  * Change in sonographic parameters; defined as score at discharge minus score at admission

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Duiverman, M.D. PhD., Study Director — University Medical Center Groningen
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided